CLINICAL TRIAL: NCT04561206
Title: A Phase 2 Study of Brentuximab Vedotin Plus Nivolumab Without Stem Cell Consolidation in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Nivolumab for the Treatment of Patients With Relapsed/Refractory Classical Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20147; NCI-2020-05332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20147 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Classic Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brentuximab vedotin, nivolumab) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Biological: Nivolumab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial investigates how well brentuximab vedotin and nivolumab work in treating patients with classical Hodgkin lymphoma that has come back after initial treatment (relapsed) or has not responded to initial treatment (refractory). Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in a targeted way and delivers vedotin to kill them. Nivolumab is an antibody that enhances the immune system to better fight Hodgkin lymphoma cells. Giving brentuximab vedotin and nivolumab may be able to defer stem cell transplant treatment and spare the considerable cost and toxicity on transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the durability of response to brentuximab vedotin (BV) plus nivolumab (nivo) by 24-month progression-free survival (PFS) in participants (with relapsed/refractory classical Hodgkin lymphoma (RcHL) after frontline therapy) who achieved early complete metabolic response (CMR) (CMR after 4 cycles).

SECONDARY OBJECTIVES:

I. Estimate CMR and overall response rate (ORR) after 4 cycles and at the end of BV-nivo therapy.

II. Estimate the PFS and overall survival (OS) for the entire cohort and for subgroups of patients defined by their response.

III. Estimate the PFS and OS separately for responders who did and did not receive radiotherapy.

IV. Evaluate the toxicities of BV-nivo in the study population.

EXPLORATORY OBJECTIVES:

I. Estimate the second PFS after salvage therapy for patients who progress after study therapy, and for the subset of these patients who proceeded to autologous stem cell transplant (ASCT).

II. Explore the association between clinical outcomes and pathological tumor characteristics.

III. Explore the association between clinical outcomes and circulating tumor deoxyribonucleic acid (ctDNA) characteristics (mutation profile, kinetics of clearance).

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes and nivolumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 16 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and 6, 12, 18, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Be willing to provide tissue (either from a fresh core or excisional biopsy performed as standard of care, or from archival tissue) of a biopsy that was performed after frontline systemic therapy, and prior to starting protocol therapy

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed diagnosis of classical Hodgkin lymphoma (excluding nodular lymphocyte predominant Hodgkin lymphoma) according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution
* Relapsed or refractory disease after no more than 1 line of prior therapy (not counting radiotherapy). However, a maximum of 5 patients with primary refractory disease may be enrolled in this study.

Note: Patients who received BV or an anti-PD-1/PD-L1 agent as part of frontline therapy are eligible if they achieved a CMR with frontline therapy and have not relapsed within 6 months from the end of frontline therapy Relapse must have been confirmed histologically (with hematopathology review at the participating institution)

* Not a candidate for ASCT, based on age, co-morbidities, or patient preference. The reason for ASCT non-candidacy must be documented in the Case Report Form and verified by the site PI
* Measurable disease (at least one non-bony fludeoxyglucose F-18 [FDG]-avid lesion >= 1.5 cm in long axis)
* Absolute neutrophil count (ANC) >= 1,000/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 50,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin >= 8 g/dL (no transfusion allowed within 3 days prior to screening)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or direct bilirubin =< 1.5 x ULN for patients with Gilbert's disease
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance of >= 40 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by women and men of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 5 months (women) or 7 months (men) after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Concomitant investigational therapy
* Live vaccine within 30 days prior to day 1 of protocol therapy (e.g. measles, mumps, rubella, varicella, yellow fever, rabies, bacillus Calmette-Guerin [BCG], oral polio vaccine, and oral typhoid)
* Grade >= 2 peripheral neuropathy
* History of prior >= grade 3 hypersensitivity to either brentuximab vedotin or nivolumab
* Known active central nervous system (CNS) involvement by lymphoma, including parenchymal and/or lymphomatous meningitis
* History of another primary malignancy that has not been in remission for at least 3 years, with the following exceptions:

  * Non-melanoma skin cancer treated with curative intent
  * In situ cervical cancer
  * If the malignancy is expected to not require any treatment for at least 2 years (this exception should be discussed with the study PI)
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration. Exceptions are:

  * Inhaled or topical steroids and
  * Adrenal replacement doses > 10 mg daily prednisone equivalents in the absence of active autoimmune disease
* History of progressive multifocal leukoencephalopathy (PML)
* Prior diagnosis of inherited or acquired immunodeficiency
* Active pneumonitis or interstitial lung disease
* Active, known or suspected autoimmune disease. The following are exceptions:

  * Vitiligo
  * Psoriasis not requiring systemic treatment
  * Hemolytic anemia associated with the lymphoma
  * Type I diabetes mellitus, if adequately controlled with therapy
  * Thyroid disease, if adequately controlled with therapy
  * Conditions not expected to recur in the absence of an external trigger (such exceptions should be discussed with the study PI)
* Active history of:

  * Hepatitis B (hepatitis B virus [HBV]) or C (hepatitis C virus [HCV]) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV DNA is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
  * Human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable human immunodeficiency virus (HIV) viral load with CD4 >= 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* History of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association class III-IV within 6 months prior to day 1 of protocol therapy
* Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 24 months in patients who achieve complete metabolic response (CMR) after 4 cycles of treatment | From start of protocol treatment to time of disease relapse/progression or death due to any cause, assessed at 24 months
  Estimated using Kaplan-Meier product limit method.

SECONDARY OUTCOMES:
Complete metabolic response (CMR) rate | After 4 or 8 cycles (each cycle is 21 days)
  Defined as the proportion of response-evaluable participants that achieve a best response of CMR with brentuximab vedotin (BV)-nivolumab (Nivo) therapy. Will be estimated along with the 95% exact binomial confidence interval.
Overall response rate (ORR) | After 4 or 8 cycles (each cycle is 21 days)
  defined as the proportion of response-evaluable participants that achieve a best response of either CMR or partial metabolic remission (PMR) with BV-Nivo therapy. Will be estimated along with the 95% exact binomial confidence interval.
Overall survival (OS) | From start of protocol treatment to time of death due to any cause, assessed up to 5 years (each cycle is 21 days)
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS/OS will be estimated when available. PFS and OS will be estimated for the entire cohort, for subgroups defined by response, and for responders who did and did not receive radiotherapy.
PFS | From start of protocol treatment to time of disease relapse/progression or death due to any cause, whichever occurs earlier, assessed up to 5 years(each cycle is 21 days)
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS/OS will be estimated when available. PFS and OS will be estimated for the entire cohort, for subgroups defined by response, and for responders who did and did not receive radiotherapy.
Incidence of adverse events | Up to 30 days post-treatment
  Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Observed toxicities of BV-Nivo therapy will be summarized by type (organ affected or laboratory determination such as absolute neutrophil count), severity, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center/John Theurer Cancer Center, Hackensack, New Jersey
  - Sarah Cannon Research Institute, Nashville, Tennessee